CLINICAL TRIAL: NCT05231980
Title: Evaluation of the Effect of Pentoxifylline and α-Lipoic Acid as Adjunctive Therapy in Patients With Clomiphene Citrate Resistant Polycystic Ovary Syndrome
Brief Title: Efficacy of Pentoxifylline and Alpha Lipoic Acid in PCOS Resistant to Clomiphene Citrate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Ahmed Abbas Morsy Morsy, principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 86
Record Dates: First submitted 2022-01-31; First posted 2022-02-09 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Clomiphene Citrate; Resistant Ovary Syndrome; Polycystic Ovary Syndrome
Keywords: pentoxifylline; alpha lipoic acid; polycystic ovary; clomiphene
MeSH Terms: conditions — Primary Ovarian Insufficiency; Polycystic Ovary Syndrome | interventions — Thioctic Acid; Pentoxifylline; Clomiphene

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pentoxifylline (PTX) group (Experimental): 30 patients
  Interventions: Drug: Pentoxifylline (PTX); Drug: Clomiphene Citrate
- Alpha lipoic acid (ALA) group (Experimental): 30 patients
  Interventions: Dietary Supplement: Alpha lipoic acid (ALA); Drug: Clomiphene Citrate
- Combined PTX and ALA group (Experimental): 30 patients
  Interventions: Dietary Supplement: Alpha lipoic acid (ALA); Drug: Pentoxifylline (PTX); Drug: Clomiphene Citrate
- control group (Active Comparator): clomiphene
  Interventions: Drug: Clomiphene Citrate

INTERVENTIONS:
Dietary Supplement: Alpha lipoic acid (ALA) — ALA is sold as a dietary supplement, either by itself or incorporated into a multivitamin product. it also has anti-oxidant effect.
  Other Names: thiotacid
  Arms: Alpha lipoic acid (ALA) group; Combined PTX and ALA group
Drug: Pentoxifylline (PTX) — Pentoxifylline is a methylxanthine derivative which acts as a vasodilator by increasing blood flow to tissues, inhibits inflammatory responses, and reduces blood viscosity by impeding platelet aggregation
  Other Names: trental
  Arms: Combined PTX and ALA group; Pentoxifylline (PTX) group
Drug: Clomiphene Citrate — is a medication used to treat infertility in women who do not ovulate
  Other Names: clomid

SUMMARY:
This study evaluate the addition of PTX and ALA to clomiphene citrate in the treatment of polycystic ovary.

DETAILED DESCRIPTION:
Clomiphene, PTX and ALA each used in treatment of pco but they do so by different mechanisms.

Clomifene is in the selective estrogen receptor modulator (SERM) family of medication. It works by causing the release of gonadotropin-releasing hormone by the hypothalamus, and subsequently gonadotropin from the anterior pituitary.

PTX and ALA are used in treatment of pco due its anti-oxidant effect.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will be diagnosed as having PCOS according to the Rotterdam criteria for diagnosis of PCOS
2. Age between 18 and 39 years.
3. Period of infertility >1 years.
4. Patients who have previously received clomiphene citrate (CC) and being diagnosed as having CC resistance
5. Body mass index (18-30) kg/m2.

Exclusion Criteria:

1. History of pelvic surgery or infertility factor other than anovulation
2. Endocrine disorders in the form of hypothyroidism or hyperthyroidism, hyperprolactinemia, and Cushing syndrome, as detected by history, examination, or investigations.
3. Known cases of endometriosis (approved histologically), uterine anomaly or hydrosalpinx, retinitis pigmentosa and vitamin K deficiency.
4. Consumption of vitamin and antioxidant supplementations in the last three-months before the trial start date.
5. Male factor infertility (sperm count < 5 million per milliliter, normal morphology <4%).
6. Elevated serum prolactin, T.S.H and F.S.H.
7. Patients diagnosed with diabetes mellitus
8. Patients who are hypersensitive to pentoxifylline or other xanthines such as caffeine, theophylline and theobromine or to any ingredient in the formulation or component of the container.
9. Patients with acute myocardial infraction, severe coronary artery disease.
10. Patients with hemorrhage or at risk of increased bleeding and Patients with peptic ulcers.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2022-06-05 (Actual); Primary Completion 2023-05-06 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
ovulation rate measure the number of patients who ovulate per cycle | 3 months
  Follicles measure more than 18 mm will be considered mature follicles.

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa Al Sabri, Phd, Study Director — Ainshams university
Locations (3):
- Egypt (3):
  - Medical Center of Infertility, Banī Suwayf
  - College of Pharmacy Teaching Hospital Ainshams University, Cairo
  - Misr University For Sciences and Technology Teaching Hospital, Giza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morsy AA, Sabri NA, Mourad AM, Mojahed EM, Fahmy SF. New insights into pentoxifylline and alpha-lipoic acid: Co-administration with clomiphene citrate for ovulation induction in anovulatory women with polycystic ovary syndrome. Clin Exp Reprod Med. 2025 May 20. doi: 10.5653/cerm.2024.07346. Online ahead of print. PMID 40393653